CLINICAL TRIAL: NCT00738881
Title: MARVEL: Marker Validation of Erlotinib in Lung Cancer- A Phase III Biomarker Validation Study of Second-Line Therapy in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Randomized to Pemetrexed Versus Erlotinib
Brief Title: Pemetrexed Disodium or Erlotinib Hydrochloride as Second-Line Therapy in Treating Patients With Advanced Non-small Cell Lung Cancer
Acronym: MARVEL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00663; NCI-2009-00663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000612010; NCCTG-N0723; CALGB-30802; CAN-NCIC-BRC4; N0723 (Other: Alliance for Clinical Trials in Oncology); N0723 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2014-12

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Pemetrexed

ARMS (2):
- Arm I (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride
- Arm II (pemetrexed disodium) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
  Arms: Arm I (erlotinib hydrochloride)
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
  Arms: Arm II (pemetrexed disodium)

SUMMARY:
This randomized phase III trial studies pemetrexed disodium to see how well it works compared with erlotinib hydrochloride as second-line therapy in treating patients with non-small cell lung cancer that has spread to other places in the body. Pemetrexed disodium and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether pemetrexed disodium is more effective than erlotinib hydrochloride in treating advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether there are differences in progression-free survival due to treatment with erlotinib (erlotinib hydrochloride) compared to pemetrexed (pemetrexed disodium) for subsets of previously treated non-small cell lung cancer (NSCLC) patients defined by epidermal growth factor receptor (EGFR)-fluorescent in situ hybridization (FISH) positive versus negativity.

SECONDARY OBJECTIVES:

I. Ascertain the presence or absence of true differences due to treatment in the objective clinical endpoints of overall survival, confirmed response rate, and adverse event profile for subsets of patients defined on the basis of the epidermal growth factor receptor (EGFR)-FISH positivity versus negativity.

II. Ascertain the presence or absence of true differences due to treatment in objective clinical endpoints (i.e., progression free survival, overall survival, confirmed response rate, and adverse event profile) for subsets of patients defined on the basis of the epidermal growth factor receptor (EGFR) expression as measured by immunohistochemistry (IHC).

III. Ascertain the presence or absence of true differences due to treatment in objective clinical endpoints (i.e., progression free survival, overall survival, confirmed response rate, and adverse event profile) for subsets of patients defined on the basis of the epidermal growth factor receptor (EGFR) gene mutation status (MUT).

IV. To evaluate the prognostic effect of EGFR copy number as measured by FISH separately by treatment arm, i.e., is there a difference in outcome for FISH(+) patients receiving erlotinib compared to FISH (-) patients receiving erlotinib, and similarly is there a difference in outcome for FISH(+) patients receiving pemetrexed compared to FISH (-) patients receiving pemetrexed.

V. To evaluate the prognostic effect of EGFR expression as measured by IHC separately by treatment arm, i.e., is there a difference in outcome for IHC(+) patients receiving erlotinib compared to IHC (-) patients receiving erlotinib, and similarly is there a difference in outcome for IHC(+) patients receiving pemetrexed compared to IHC (-)patients receiving pemetrexed.

VI. To evaluate the prognostic effect of EGFR mutation status separately by treatment arm, i.e., is there a difference in outcome for MUT(+) patients receiving erlotinib compared to MUT(-) patients receiving erlotinib, and similarly is there a difference in outcome for MUT(+) patients receiving pemetrexed compared to MUT(-) patients receiving pemetrexed.

VII. To prospectively test the hypothesis that functionally relevant polymorphisms in the genes encoding for pemetrexed targets, as well as genes encoding for one or more of the key enzymes involved in the transport, activation, and inactivation of pemetrexed, either singly or in combination, play a role in the efficacy and/or toxicity of pemetrexed.

VIII. To prospectively test the hypothesis that functionally relevant polymorphisms in the EGFR gene as well as genes encoding for one or more of the key enzymes involved in the metabolism of erlotinib, either singly or in combination, play a role in the efficacy and/or toxicity of erlotinib.

IX. Evaluate proteomic signatures in blood samples as predictors of survival and response to treatment with erlotinib.

X. To evaluate expression of thymidylate synthase, dihydrofolate reductase, phosphoribosylglycineamide (GAR) formyltransferase, and methylthioadenosine phosphorylase gene expression in tumor samples, as measured by IHC or quantitative polymerase chain reaction, as predictors of survival and response to treatment with pemetrexed.

XI. To evaluate proteomic signatures in blood samples of patients as predictors of response and survival to treatment with erlotinib.

XII. To evaluate the following variables measured in tumor samples, as predictors of response and survival to treatment with pemetrexed: Expression of thymidylate synthase, dihydrofolate reductase and GAR formyltransferase genes methylthioadenosine phosphorylase expression by IHC or quantitative polymerase chain reaction (PCR).

XIII. To evaluate the following variables measured in tumor samples, as predictors of response and survival to treatment with erlotinib: Rat sarcoma (Ras) mutational status, EGFR mutational status and, epithelial to mesenchymal transition (EMT) status (measured by E-cadherin expression and vimentin expression) by IHC.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pemetrexed disodium intravenously (IV) over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented recurrence or disease progression of NSCLC

  * NSCLC must be confirmed by pathologic examination, either on initial diagnosis or disease recurrence/progression; mixed histology allowed if all components consistent with NSCLC
* Measurable disease, defined as at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm by conventional techniques or as >= 1.0 cm by spiral computed tomography (CT); if spiral CT is used, it must be used for both pre- and post- treatment tumor assessments
* Prior radiation therapy is permitted as long as:

  * Recovered from the toxic effects of radiation treatment before study entry, except for alopecia
  * =< 25% of bone marrow radiated
  * Presence of measurable disease whether in-field disease progression/recurrence or disease outside the treatment fields of radiation port
* Absolute neutrophil count (ANC) >= 1,500 uL
* Platelet (PLT) >= 100,000 uL
* Hemoglobin (Hgb) >= 10 g/dL
* Total bilirubin: within normal institutional limits (WNL) OR direct bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* International normalized ratio (INR) =< 1.5
* Calculated creatinine clearance >= 45 mL/min using the Cockcroft-Gault formula
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Negative pregnancy test done =< 7 days prior to pre-registration, for women of childbearing potential only
* Ability to provide informed consent
* Life expectancy >= 12 weeks
* Tissue available and willing to submit tissue for central pathology review and EGFR evaluation; performed on original diagnostic/recurrent tissue (preferably paraffin-embedded tissue blocks); if institution unable to release tissue blocks, willing to submit 25 unstained slides (15 sections cut at 5 microns mounted on charged slides and 10 sections cut at 10 microns mounted on uncharged slides)
* Must be previously treated for advanced disease with only 1 chemotherapy regimen which must contain cytotoxic agent(s); adjuvant/neoadjuvant treatment with cytotoxic agent(s) administered < 12 months (from date chemotherapy was started) prior to pre-registration will be considered as one prior treatment; NOTE: adjuvant/neoadjuvant treatment administered >= 12 months, use of targeted agents such as monoclonal antibodies prior to pre-registration will NOT be counted as one prior treatment; patient could have had adjuvant/neoadjuvant chemotherapy >= 12 months and 1 systemic chemotherapy regimen for metastatic or recurrent disease
* Able to take folic acid, vitamin B12 supplementation, and dexamethasone
* Able to permanently discontinue aspirin dose of >= 1.3 grams/day >= 10 days before and after pemetrexed treatment
* Fertile patients must use effective contraception
* Able to take folic acid, vitamin B_12 supplementation, and dexamethasone
* Stable brain metastasis that have been treated with either whole brain radiation therapy or gamma knife surgery and are off steroid treatment for > 14 days prior to pre-registration, if applicable
* Willingness to return to enrolling institution for treatment and follow-up

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any clinically significant infection, at the treating physician's discretion
* Known human immunodeficiency virus (HIV) positive patients
* Impairment of gastrointestinal (GI) function, inability to swallow pills in the absence of a feeding tube, or GI disease that may significantly alter absorption of oral medications (e.g. ulcerative disease, uncontrolled nausea and vomiting, malabsorption syndromes, bowel obstruction, etc)
* Serious condition that, in the opinion of the investigator, would compromise the patient's ability to complete the study or increase the risk for serious adverse events
* Any of the following prior therapies:

  * Prior radiation to > 25% of bone marrow
  * EGFR tyrosine kinase inhibitors
  * Pemetrexed
  * Chemotherapy =< 3 weeks prior to pre-registration
  * Mitomycin C/nitrosoureas =< 6 weeks prior to pre-registration
  * Immunotherapy =< 2 weeks prior to pre-registration
  * Biologic therapy =< 2 weeks prior to pre-registration
  * Gene therapy =< 2 weeks prior to pre-registration
  * Full field radiation therapy =< 4 weeks prior to pre-registration
  * Limited field radiation therapy =< 2 weeks prior to pre-registration
  * Major surgery (i.e., laparotomy), open biopsy, or significant traumatic injury =< 4 weeks prior to pre-registration or anticipation of need for major surgical procedure during the course of the study; minor surgery =< 2 weeks prior to pre-registration; insertion of a vascular access device is not considered major or minor surgery in this regard
* Other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) =< 4 weeks prior to pre-registration
* Steroid therapy for brain metastasis =< 14 days prior to pre-registration
* Symptomatic serosal effusion (>= Common Terminology Criteria for Adverse Events [CTCAE] v3.0 grade 2 dyspnea) that is not amenable to drainage prior to pre-registration
* Other invasive solid or hematologic malignancy; exceptions: prior malignancy was diagnosed and definitively treated >= 5 years previously with no subsequent evidence of recurrence; patients with a history of low-grade (Gleason score =< 6) localized prostate cancer will be eligible even if diagnosed < 3 years prior to pre-registration; these patients may continue on medications concomitantly to maintain their disease remission as necessary; patients with carcinoma in situ, regardless of organ involvement, or non-melanoma cutaneous carcinomas are eligible if these were definitively treated >= 3 years previously with no subsequent evidence of recurrence; Note: patients with breast cancer that was definitively treated > 5 years earlier but continue to receive aromatase inhibitors are NOT eligible
* Only non-measurable disease, defined as all other lesions, including small lesions whose longest diameter measures < 2 cm with conventional techniques or < 1.0 cm with spiral CT, and truly non-measurable lesions, which include the following as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria dated June 1999:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Single disease site in prior radiation field
* Any of the following concurrent severe and/or uncontrolled medical conditions:

  * Angina pectoris
  * History of congestive heart failure =< 3 months prior to pre-registration, unless ejection fraction > 40%
  * Myocardial infarction =< 6 months prior to pre-registration
  * Cardiac arrhythmia
  * Diabetes mellitus
  * Hypertension
  * Any other severe underlying diseases which are, in the judgment of the investigator, inappropriate for entry into this study
* Respiratory symptoms > CTCAE grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (269):
- United States (268):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Bristol Hospital, Bristol, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Cancer Trials Support Unit, Rockville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Minnesota Cooperative Group Outreach Program, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Cancer Consortium-Upstate NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty nine (29) pre-registered, screen failures (4 inadequate tissue, 1 investigator decision and one patient decision). Twenty three (23) patients were randomized, 2 patients withdrew from study prior to receiving any study treatment, thus a total of 23 randomized patients are evaluable for the primary and secondary endpoints.
Groups:
- Arm I: Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given orally
- Arm II: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  pemetrexed disodium: Given IV
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 11 | 12
Completed | 11 | 10
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 76] | 55 [49 to 75] | 62 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated using the method of Kaplan-Meier survival curves to compare PFS between the erlotinib and pemetrexed arms using an intent-to-treat (ITT) analysis. Due to the small sample size (21 of the required 954 patients ~2%), analyses within the FISH(+) and FISH(-) groups were not performed, and no formal analyses for the primary or the secondary efficacy outcomes were performed.
Time Frame: Time from randomization to the first date of documented disease progression or death, assessed up to 5 years
Population: All the 23 randomized patients are eligible for primary end point analysis using an ITT principle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 11 | 12
months | 2 [1.3 to 6.9] | 3.1 [1.2 to 4.2]

2. Secondary Outcome: Time to Treatment Failure
Description: The distribution of all time to event data will be estimated using the method of Kaplan-Meier survival curves.
Time Frame: The time from date of randomization to the date at which the patient is removed from the treatment, assessed up to 5 years
Population: Since the trial closed prematurely with only ~2% accrual, the secondary outcomes were not analyzed.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan-Meier survival curves. A 1-sided stratified log rank test [accounting for all the stratification factors except FISH status and cooperative group] will be used to compare overall survival between the erlotinib and pemetrexed arms within the FISH(+) and FISH(-) subgroups, compare overall and progression free survival between the erlotinib and pemetrexed arms within the subgroups defined on the basis of the epidermal growth factor receptor (EGFR) expression by immunohistochemistry (IHC), and EGFR gene mutation status (MUT). Cox proportional hazards model will be used to assess potential differences.
Time Frame: Time from randomization to time of death from any cause, assessed up to 5 years
Population: Since the trial closed prematurely with only ~2% accrual, the secondary outcomes were not analyzed.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Confirmed Response Rate Defined as Complete Response (CR) or a Partial Response (PR) Per Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. The proportion of patients with confirmed CR and PR will be computed within each treatment arm and exact binomial confidence intervals for the true proportion computed. Chi-square test and Fisher's exact test will be used to compare the response rates between the treatment arms within the subgroups defined by FISH status, IHC, and MUT.
Time Frame: Up to 5 years
Population: Since the trial closed prematurely with only ~2% accrual, the secondary outcomes were not analyzed.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm I: erlotinib hydrochloride: Given orally
- Arm II: pemetrexed disodium: Given IV
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=11) | Arm II (N=10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (24) | 8 (30)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 3 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 4 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 9 (49) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (17) | 6 (15)
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 (4)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (49) | 10 (38)
Fever (General disorders) | 1 (1) | 4 (7)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (13) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 2 (3)
Bilirubin increased (Investigations) | 3 (4) | 0 (0)
Creatinine increased (Investigations) | 3 (4) | 2 (3)
Leukocyte count decreased (Investigations) | 4 (20) | 2 (5)
Lymphocyte count decreased (Investigations) | 1 (4) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (5)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 4 (8) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 7 (19) | 6 (14)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 9 (25)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (47) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (23) | 2 (3)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less